CLINICAL TRIAL: NCT01625624
Title: Effect of Food Products on Perceived Energy and Task Performance
Brief Title: Evaluating the Effects of Food Products on Energy and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KFG-122X-02
Record Dates: First submitted 2012-06-05; First posted 2012-06-21 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Energy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Food Product (Placebo Comparator)
  Interventions: Other: Carbohydrate Food Bar
- Experimental Food Product (Experimental)
  Interventions: Other: Modified Carbohydrate Food Bar

INTERVENTIONS:
Other: Carbohydrate Food Bar — Control Food Bar containing carbohydrate
  Arms: Control Food Product
Other: Modified Carbohydrate Food Bar — Test Food Bar containing modified carbohydrate
  Arms: Experimental Food Product

SUMMARY:
The purpose of this study is to determine the effect of food products varying in composition, on energy in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 years (inclusive).
* English as primary language.
* Have a minimum of a high school degree (note that GED is not sufficient).
* Females of Child-bearing Potential (FOCP) must have a negative urine or serum beta HCG pregnancy test at screening. FOCP must abstain from sexual activity that could result in a pregnancy, or use acceptable contraceptives throughout the period of study treatment exposure and for 30 days after the last study treatment. Acceptable contraceptives include IUDs, hormonal contraceptives (oral, implanted or injectable) and double barrier methods (such as condom or diaphragm with spermicidal gel). If hormonal contraceptives are used, the period of use must be sufficiently long to achieve pharmacological effectiveness prior to study treatment exposure (refer to individual product information for details on onset of effectiveness). FOCP who are not currently sexually active, must agree to use acceptable contraception, as defined above, if they decide to become sexually active during the period of study treatment exposure and for thirty days thereafter.
* Good physical and mental health based on a general medical, mental health questionnaire.
* Adequate visual, auditory and cognitive ability to complete the assessments within the Normal range (i.e., no more than 1 standard deviation below the mean for the subject's age and years of education).
* Willing and able to comply with all requirements defined within this protocol.
* Willing to obtain at least 7 hours of nighttime sleep during the evenings prior to study visits.
* Willing to avoid strenuous exercise for 24 hours prior to visits.
* Willing to avoid alcohol for 24 hours prior to visits.
* Willing to abstain from caffeine after midnight prior to visits.
* Moderate daily user of caffeine (approximately 1-4 cups of coffee or equivalent per day).

Exclusion Criteria:

* Current Axis I or Axis II comorbid psychiatric diagnosis or other symptomatic manifestations that, in the opinion of the examining physician (Investigator), will contraindicate treatment with caffeine.
* Attention Deficit Hyperactivity Disorder.
* BMI ≤ 19 or ≥ 30 kg/m2.
* History of drug dependence or substance use disorder based upon DSM-IV-TR criteria (excluding nicotine).
* Positive urine drug or alcohol drug test result.
* Users of nicotine products within 30 days of screening or during the duration of the study.
* Taking any over the counter or prescription medications other than birth control.
* Concurrent chronic or acute illness (such as allergic rhinitis or severe cold), disability, or other condition that might confound the results of rating tests administered in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional conditions that, in the Investigator's opinion, would preclude the subject from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol.
* Participation in an investigational study or received an investigational drug within the past 28 days.
* Individuals who do not maintain a routine nighttime sleep schedule (no shift work).
* Pregnant or lactating women, or women planning to become pregnant during the study.
* Hypertension or other chronic medical conditions.
* Judged by the Investigator to be unsuitable for enrollment in this study for any reason.
* Has been diagnosed with phenylketonuria.
* Individuals with sleep disorders (e.g. sleep apnea, primary or secondary insomnia).
* Known pre-existing medical condition.
* Has a fasting glucose of >110 mg/dl.
* Has an allergy to wheat, soy, nuts or any other food.
* Has Kosher or Halal dietary restrictions.
* Reports never eating biscuits, cookies or crackers.
* Epworth Sleepiness Scale ≥ 12 at screening (i.e., evidence of excessive daytime sleepiness).

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Subjective feeling of energy (visual analog scale) | 150 minutes post food consumption

CONTACTS AND LOCATIONS:
Overall Officials: Gary Kay, PhD, Principal Investigator — Cognitive Research Corporation
Locations (2):
- United States (2):
  - Renstar Medical Research, Ocala, Florida
  - Cognitive Research Corporation, St. Petersburg, Florida